CLINICAL TRIAL: NCT02262494
Title: Location of Lower Extremity Deep Vein Thrombosis by Emergency Physicians Using Portable Compression Ultrasonography: a Diagnostic Study
Brief Title: Location of Lower Extremity Deep Vein Thrombosis by Emergency Physicians Using Portable Compression Ultrasonography
Acronym: EchoComp TVP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No recruitment
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2013/XB-01; 2014-A00510-47 (Other: RCB number)
Record Dates: First submitted 2014-10-02; First posted 2014-10-13 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suspected first episode of DVT (Other): The study population consists of patients presenting with suspected first episode of DVT at the Nîmes University Hospital.
  Intervention: portable venous compression ultrasonography Intervention: venous compress ultrasonography Intervention: Doppler ultrasound of the lower limbs
  Interventions: Procedure: portable venous compression ultrasonography; Procedure: venous compress ultrasonography; Procedure: Doppler ultrasound of the lower limbs

INTERVENTIONS:
Procedure: portable venous compression ultrasonography — venous compression ultrasonography performed using an ultra-portable ultrasound device (by emergency physician)
Procedure: venous compress ultrasonography — venous compression ultrasonography performed using a classic ultrasound device (by exploratory specialist)
Procedure: Doppler ultrasound of the lower limbs — Doppler ultrasound of the lower limbs (gold standard; by exploratory specialist)

SUMMARY:
The main objective of our study is to determine the diagnostic performance of an ultra-portable ultrasound (V-Scan®) device for emergency compression ultrasound when used by experienced ermergency doctors searching for proximal deep vein thrombosis (DVT) in patients with no history of DVT. The gold standard is Doppler ultrasound of the lower limbs performed by a vascular exploration expert.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* to compare the diagnostic performance of emergency compression ultrasonography performed with and ultra-portable device (V-Scan®) with that of emergency compression ultrasonography performed with a classic device
* to compare the diagnostic performance of emergency compression ultrasonography between patients suspected of having DVT arriving through the emergency department versus similar patients sent in by their generalist
* to compare the diagnostic performance of emergency compression ultrasonography among patients with suspected DVT according to pre clinical probability testing based on the Wells score (low, medium or high probability).

Currently, the use of ultra-portable ultrasound in this indication is not part of routine care, and this study is therefore considered interventional in nature.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given informed consent and signed consent
* The patient must be a member or beneficiary of a health insurance plan
* Patient consulting in the vascular exploration and medicine department for suspected first episode of deep vein thrombosis
* Ambulatory patient: defined as any outpatient coming in for a consult directly from their place of residence or via the emergency department
* Patient does not have a history of venous thromboembolism

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is an adult under any kind of guardianship
* The patient refuses to sign the consent
* It is not possible to correctly inform the patient
* Patient has a history of venous thromboembolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-10-19 (Actual)

PRIMARY OUTCOMES:
Diagnosis of deep vein thrombosis by portable ultrasound: yes/no | Day 0
Diagnosis of deep vein thrombosis by doppler ultrasound: yes/no | Day 0

SECONDARY OUTCOMES:
Diagnosis of deep vein thrombosis by classic ultrasound: yes/no | day 0
Wells score | Day 0
  score ranging from 0 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Bobbia, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France